CLINICAL TRIAL: NCT02956226
Title: Cannabinoids for Behavioral Problems in Autism Spectrum Disorder: A Double Blind, Randomized, Placebo-controlled Trial With Crossover.
Brief Title: Cannabinoids for Behavioral Problems in Children With ASD
Acronym: CBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Adi Aran, Director, Neuro-pediatric unit, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBA
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Cannabinoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cannabinoids - 99% pure cannabinoids mix (Experimental): Oral cannabinoids mix [cannabidiol (CBD), Δ9-tetrahydrocannabinol (THC) in a 20:1 ratio] at 1 mg/kg cannabidiol per day, up-titrated until intolerance or to a maximum dose of 10 mg/kg CBD per day, divided to 3 daily doses, for 3 months.
  Interventions: Drug: Cannabinoids - 99% pure cannabinoids mix
- Placebo (Placebo Comparator): Oral olive oil and flavors that mimic in texture and flavor the cannabinoids' solution.
  Interventions: Drug: Placebo
- Cannabinoids - whole plant extract (Experimental): Oral cannabinoids mix [cannabidiol (CBD), Δ9-tetrahydrocannabinol (THC) in a 20:1 ratio] at 1 mg/kg cannabidiol per day, up-titrated until intolerance or to a maximum dose of 10 mg/kg CBD per day, divided to 3 daily doses, for 3 months
  Interventions: Drug: Cannabinoids - whole plant extract

INTERVENTIONS:
Drug: Cannabinoids - 99% pure cannabinoids mix — 99% pure cannabidiol (CBD) and 99% pure Δ9-tetrahydrocannabinol (THC) in a 20:1 ratio (B.O.L Pharma, Israel), in a 160/8.0 mg per mL (CBD/THC) olive oil-based solution.
  Arms: Cannabinoids - 99% pure cannabinoids mix
Drug: Placebo — Olive oil and flavors solution.
  Arms: Placebo
Drug: Cannabinoids - whole plant extract — Whole plant extract enriched with cannabidiol (CBD) and Δ9-tetrahydrocannabinol (THC) to achieve 20:1 ratio (B.O.L Pharma, Israel), in a 160/8.0 mg per mL (CBD/THC) olive oil-based solution.
  Arms: Cannabinoids - whole plant extract

SUMMARY:
This study aims to assess the safety, tolerability and efficacy of cannabinoids mix [cannabidiol (CBD), Δ9-tetrahydrocannabinol (THC) in a 20:1 ratio, BOL Pharma, Israel] for behavioral problems in children and youth with ASD.

DETAILED DESCRIPTION:
Disruptive behaviors are very common in children and youth with autism spectrum disorder (ASD). Behavioral problems increase social impairment in children with ASD, make interventions more difficult and place considerable strain on families and caregivers. Current treatment is based on behavioral interventions combined with atypical antipsychotics which often have low tolerability and questionable efficacy.

Cannabis exerts profound effects on human social behavior. Research using animal models of ASD indicate a possible dysregulation of the endocannabinoid system, and stress that it may be a novel target for pharmacological interventions. Anecdotal evidence suggest efficacy of various phytocannabinoids in resistant behavioral problems. However controlled human studies are lacking.

Objective: To assess the safety, tolerability and efficacy of cannabinoids mix [cannabidiol (CBD), Δ9-tetrahydrocannabinol (THC) in a 20:1 ratio, BOL Pharma, Israel] for behavioral problems in children and youth with ASD.

Setting: A double blind randomized placebo-controlled trial with crossover.

Methods: One hundred and fifty participants, ages 5-21 years, with ASD and moderate to severe refractory behavioral problems will be randomized to receive 1 out of 3 treatments for 12-weeks and cross-over to another treatment in a second 12 weeks period. Treatment options are: (1) oral placebo (2) cannabis extract, contains cannabidiol and Δ9-tetrahydrocannabinol in a 20:1 ratio, at a cannabidiol dose of 10 mg/kg/d and (3) pure cannabidiol and Δ9-tetrahydrocannabinol in the same ratio and dose.

Outcomes and measures: Two co-primary endpoints will compare the whole plant extract treatment to the placebo treatment on a within subject design. 1) The change from baseline Home Situations Questionnaire-ASD score after 3 months of treatment (HSQ-ASD; a parent rated assessment of disruptive behavior). 2) The Clinical Global Impression- improvement (CGI-I; a clinician rated assessment of improvement in disruptive behavior following treatment)

Secondary efficacy outcomes include:

* Within subject differences between the placebo condition and the pure cannabinoids condition and between the whole plant extract condition and the pure cannabinoids condition in the change from baseline HSQ-ASD score after 3 months of treatment and in the CGI-I.
* Within subject differences between each pair of the 3 conditions in the Clinical Global Impression- drug effect (CGI-D).
* Within subject differences between each pair of the 3 conditions in the change from baseline after 3 months of treatment in: Social Responsiveness Scale (SRS) parent and teacher rated, Child Behavior Checklist (CBCL) and autism parenting stress index (APSI).

Safety endpoints will include the proportion of patients with adverse events measured by the investigators and the Liverpool Adverse Events Profile (modified).

Exploratory measures are: markers of the endocannabinoid system in the patients' blood and possible correlation to phytocannabinoids bioavailability and treatment response, change from baseline at the end of treatment in BMI and Children's Sleep Habits Questionnaire (CSHQ) score and quality of parent- child interaction during the study (Emotional Availability- EA).

Long term safety, tolerability and efficacy of cannabidiol-rich medical cannabis will be assessed after 12 and 24 months of open treatment, in a subgroup of patients who will apply for medical license to use cannabis after completing the study.

ELIGIBILITY:
Inclusion Criteria: (both are needed)

* ASD diagnosis (Diagnostic and Statistical Manual of Mental Disorders [Fifth Edition; DSM-V]
* Moderate or greater behavioral problems as measured by a rating of moderate or higher (≥4) on the Clinical Global Impression-Severity (CGI-S)

Exclusion Criteria:

* Planned changes in existing interventions for the duration of the trial or such a change in the last 4 weeks.
* Current treatment with cannabis based therapy or such a treatment in the last 3 months.
* Heart, liver, renal or hematological disorders
* History of psychotic disorder in a first degree relative.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Home Situations Questionnaire-Autism Spectrum Disorder (HSQ-ASD) score, at three months. Within subject difference between the placebo condition and the whole plant extract condition. | At onset of each treatment period, at 1 month, 2 months and 3 months (end of treatment period)
  This is a 24-item parent-rated measure of noncompliant behavior in children with ASD
Clinical Global Impression-Improvement scores (CGI-I ) at three months. Within subject difference between the placebo condition and the whole plant extract condition. | At 3 months (end of treatment period)
  This is a 7-point scale designed to measure overall improvement from baseline (CGI-I).

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement scores (CGI-I ) at three months. Within subject differences between the placebo condition and the pure cannabinoids condition and between the whole plant extract condition and the pure cannabinoids condition. | At 3 months (end of treatment period)
  This is a 7-point scale designed to measure overall improvement from baseline
Change in Social Responsiveness Scale scores-2 (SRS-2, parent and teacher rated) at three months | At onset of each treatment period and at 3 months (end of treatment period)
  This is a 65 item, caregiver (pSRS) or teacher (tSRS) questionnaire, used to determine the severity of social deficit exhibited by participants with ASD. The SRS contains five subscales: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Autistic Mannerisms, which respectively measure the ability to recognize social cues, the ability to interpret social cues, the ability to use expressive verbal and nonverbal language skills, the ability to engage in social-interpersonal behaviors, and the tendency to display stereotypical behaviors and restricted interests characteristic of autism
Change in Autism Parenting Stress Index (APSI) score, at three months | At onset of each treatment period, at 1 month, 2 months and 3 months (end of treatment period)
  This is a 13-item parent rated measure designed to assess the effect of interventions to control disruptive behavior in children with ASD on parenting stress.
Change from baseline Home Situations Questionnaire-Autism Spectrum Disorder (HSQ-ASD) score, at three months. | At onset of each treatment period, at 1 month, 2 months and 3 months (end of treatment period)
  This is a 24-item parent-rated measure of noncompliant behavior in children with ASD. Within subject differences between the placebo condition and the pure cannabinoids condition and between the whole plant extract condition and the pure cannabinoids condition.

OTHER OUTCOMES:
Modified Liverpool Adverse Events Profile (LAEP) | At onset of each treatment period, at 1 month, 2 months and 3 months (end of treatment period)
  Tolerability and adverse effects will be assessed using this modified Liverpool Adverse Events Profile (LAEP) that includes all 19 items of the original LAEP and another 15 items to cover all reported significant side effects of CBD and THC in former studies.

CONTACTS AND LOCATIONS:
Overall Officials: Adi Aran, MD, Principal Investigator — Shaare Zedek Medical Center; Varda Gross, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aran A, Harel M, Cassuto H, Polyansky L, Schnapp A, Wattad N, Shmueli D, Golan D, Castellanos FX. Cannabinoid treatment for autism: a proof-of-concept randomized trial. Mol Autism. 2021 Feb 3;12(1):6. doi: 10.1186/s13229-021-00420-2. PMID 33536055